CLINICAL TRIAL: NCT00736463
Title: Effects of High Dose Simvastatin vs. Atorvastatin on Baseline Lipoprotein Profiles, Apo-A-1 and C Reactive Protein
Brief Title: Crossover of Higher Dose Statins in Patients With Low High-density Lipoproteins Cholesterol (HDLc)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Oregon State University (Other); Indiana University (Other)
Responsible Party: Craig D. Williams, Pharm.D. Clinical Associate Professor, OHSU/OSU School of Pharmacy
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00004506
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-08

CONDITIONS: HDL Cholesterol
Keywords: HDL cholesterol; statin; inflammation; atherosclerosis; prevention; patients with low baseline HDL cholesterol
MeSH Terms: conditions — Inflammation; Atherosclerosis | interventions — Simvastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Aimvastatin 80 mg
  Interventions: Drug: Simvastatin
- 2 (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin 80 mg

INTERVENTIONS:
Drug: Simvastatin — One arm of randomized crossover
  Arms: 1
Drug: Atorvastatin 80 mg — Second arm of randomized crossover
  Arms: 2

SUMMARY:
Summary:

Background: There is a lot of interest in the function and role of HDL to prevent and mitigate atherosclerosis in patients who are at or near LDLc targets. Statins have variable effects on HDLc which are accentuated in patients with a low baseline HDLc. Higher doses of statins are being used more commonly in practice based on newer outcomes studies which find greater benefits of the higher doses compared to lower or standard doses. This study is testing FDA approved dosages of two commonly used statin medications.

Design: The study is designed to examine the effects of 80mg simvastatin and 80mg atorvastatin on HDLc concentrations. Serum will be saved for a hopeful collaborative effort with investigators at the U. of Washington who are able to do more advanced testing of HDL particle functionality. Based on the first 13 patients studied at Indiana University, the effects of these statins on HDLc concentrations vary greatly. It is unknown what impact these concentration changes have on the functionality of the particles however. A meta-analysis of 4 prospective trials published in JAMA in 2006 found that increasing HDLc with statins was independently associated with regression of atherosclerosis as measured by intravascular ultrasound.

Patients: Patients with low HDLc will be the primary population recruited. Exclusion criteria include interacting medications, pregnancy, baseline hepatic disease or other illnesses which would put patients at increased risk of statin side effects.

DETAILED DESCRIPTION:
The subject will be asked to come in for all study visits in a fasting state (only water for past 12 hours). Both blood pressure and pulse will be checked at the screening visit as well as all study visits. The baseline (screening) visit will include the consenting process and completion of the first section of the Data Collection Sheet to further screen for appropriate inclusion and exclusion criteria. Subjects who are on a statin will need to have an 8-week wash out period prior to beginning the trial. The subject and their primary provider must agree to the washout.

At the screening visit for subjects not taking a statin drug, 13 ml of blood will be drawn. The blood will be processed by the OCTRI Core Laboratory staff. All of the lipid parameters (complete lipid profile, apoB, apoA1, hs-CRP) will be tested at the OHSU lipid core lab. Some of the blood collected will be sent to the OHSU core lab for testing of ALT as well as for obtaining the long-term storage sample. Blood samples will be frozen and stored on the 14th floor of the CHH building in the laboratory of the Oregon State University School of Pharmacy. Samples will be batched for processing (see sample processing below). The lipid profile and ALT from the screening visit will be processed within approximately one week. If necessary laboratory parameters meet inclusion and exclusion criteria, the subject will be scheduled for the first study visit. Encapsulated placebo will be given to the subject to take in between the screening and first study visit.

At the screening visit for subjects taking a statin drug, the study will be described and consent to enroll will be obtained but no bloodwork will be performed. Subjects will be given an encapsulated placebo to take for an 8 week washout period. At the second screening visit, blood will be drawn to ascertain baseline laboratory values as described above for subjects not on a statin drug. The subject will then be scheduled for their first study visit 2 weeks later.

The other laboratory parameters (hs-CRP, apoA1 and apoB) and all future bloodwork which is not necessary for the ongoing conduct of the trial may be batched and processed periodically. The ALT from the second study visit (after first course of study medication) will be processed prior to the third study visit to confirm that ALT remains less than 3 times ULR. If ALT is elevated (>105 IU/L) at the second study visit, the subject will be discontinued from the study and the subjects primary physician notified. Additionally, if the subject complains of myopathy which is felt to be consistent with possible drug-induced myositis, a creatine phospho-kinase (CPK) test will be ordered. Consistent with the product package insert (PI) for both atorvastatin and simvastatin, therapy will be stopped and the subject discontinued from the study if CPK is greater than 10X the ULR.

At the first study visit, the subject will be randomized by the OHSU Research Pharmacy to receive either 6 weeks of 80mg atorvastatin or 6 weeks of 80mg of simvastatin. The subject will be scheduled for follow-up 6 weeks from the trial entry date and asked to bring the investigational drug vial back at the next visit. The subjects will also be given a diary to record their daily dose of medication taken. A urine pregnancy test will be done at the first and third study visit in all women who are not post-menopausal as defined as at least 6 months without menstruation over the age of 50. Women who do not meet the post-menopausal criteria, are sexually active and not on any form of birth control will be counseled to begin and remain on birth control for the duration of the trial. Inability or unwillingness to comply with chosen birth control measures will result in exclusion from the trial. Women of child bearing potential not on birth control at the time of the screening visit who are willing to begin birth control will be scheduled for their first study visit not sooner than 6 weeks after their screening visit to allow time for implementation of chosen birth control. Subjects who are on hormone replacement therapy (HRT) will be allowed to enroll provided that their regimen is stable and not expected to change during the study period. Subjects will be informed that if their regimen does change during the study, they will need to be removed from the study.

At the second visit, the appropriate section of the Data Collection Sheet will be completed, a pill count of remaining drug doses will be done and 13 ml of blood will be drawn and processed as previously outlined. The subject will then be scheduled for follow-up in 6 weeks and leave without any study medicine.

At the third visit, the appropriate section of the Data Collection Sheet will be completed and 13 ml of blood will be drawn and processed as previously outlined. The subject will be given a 6 week supply of the second medication (as previously determined by first randomization scheme) and scheduled for follow-up in 6 weeks.

At the fourth and final visit, the appropriate section of the data collection sheet will be completed and 13 ml of blood will be drawn and processed as previously outlined.

In between study visits, the study staff will contact subjects by phone to remind them of their next appointment and ask about any adverse effects or other problems that the subject may be experiencing. In the event that the phone number of record becomes inactive, a letter will be sent to the address of record.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Screening visit HDL-c cholesterol < 40 mg/dL (men) or < 50 mg/dL (women)
* Screening visit LDL-c or non-HDL-c (for patients with TG 200-500 mg/dL) in range requiring therapy based on National Cholesterol Education Program (NCEP) guidelines
* Identifiable primary care provider
* Working phone number for follow-up

Exclusion Criteria:

* Age < 18 years
* Any unstable coronary disease (angina) at the screening visit or any acute coronary syndrome < 6 months prior to first study visit
* Screening TG > 750 mg/dL
* Known allergy or contraindication to atorvastatin or simvastatin
* Known HIV/AIDS diagnosis
* Screening alanine aminotransferase (ALT) > 3 times upper lab reference range (ULR)
* Known history or diagnosis of clinical hepatic failure (example: variceal bleeding, ascites, INR>1.3)
* Self-reported weekly alcohol intake of > 2 drinks per day on average (e.g. > 14 drinks/week)
* Self- reported pregnancy or current breastfeeding
* Use of a fibrate or niacin product or any other drug listed in the Zocor or Lipitor product package insert at a dose which causes a significant drug interaction
* Anticipated inability to complete the 4-visit study timeline for any reason (expected prolonged travel, extenuating medical needs, etc.)
* Active participation in another research protocol which would interfere with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
HDL cholesterol | 6 weeks

SECONDARY OUTCOMES:
HS-CRP, apolipoprotein A1 and B | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Williams, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Hospital, Portland, Oregon, United States

REFERENCES:
- [Result] Deeg MA, Raikwar NS, Johnson C, Williams CD. Statin therapy reduces serum levels of glycosylphosphatidylinositol-specific phospholipase D. Transl Res. 2007 Sep;150(3):153-7. doi: 10.1016/j.trsl.2007.03.008. Epub 2007 May 25. PMID 17761367
- See also: Related Info — http://www.ohsu.edu/xd/research/index.cfm